CLINICAL TRIAL: NCT03294564
Title: Cognitive, Emotional, and Neural Responses to Acute Inflammation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14-13204; K01MH109871 (NIH)
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Healthy
Keywords: Inflammation; Threat sensitivity; Reward sensitivity
MeSH Terms: conditions — Inflammation | interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Typhoid Vi Polysaccharide Vaccine (Active Comparator): Patients will receive one intramuscular 0.5 mL injection of Typhoid Vi Polysaccharide Vaccine containing 0.025 mg purified Vi polysaccharide.
  Interventions: Biological: Typhoid Vi Polysaccharide Vaccine
- Placebo (Placebo Comparator): Patients will receive one intramuscular 0.5 mL injection of saline placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Typhoid Vi Polysaccharide Vaccine — Salmonella typhi capsular polysaccharide vaccine (Typhoid Vi Polysaccharide Vaccine): Each dose of 0.5ml Salmonella typhi capsular polysaccharide vaccine (Sanofi Pasteur, SA) is formulated to contain 25μg of purified Vi polysaccharide in a colorless isotonic phosphate buffered saline (pH 7±0.3), 4.150mg of sodium chloride, 0.065mg of disodium phosphate, 0.023mg of monosodium phosphate and 0.5ml of sterile water for injection. It is indicated for use by humans aged 2 years and older for protection against typhoid fever.
  Arms: Typhoid Vi Polysaccharide Vaccine
Biological: Placebo — The placebo injection will consist of 0.5mL of saline.
  Arms: Placebo

SUMMARY:
This study is a pilot study to examine the effects of acute inflammation on cognition and emotion in healthy participants using a between-subjects, randomized, double-blind design.

DETAILED DESCRIPTION:
The inflammatory response of the immune system is responsive to stress and it impacts brain function. Animal studies have shown that inflammation appears to alter threat- and reward-related brain activity. Accumulating evidence points to inflammatory proteins, specifically cytokines, as key players in this relationship. Although cytokines are typically too large to pass through the blood brain barrier (BBB), they can influence brain function and structure by transmitting signals from peripheral systems to the brain.

The administration of endotoxin within the polysaccharide form of Salmonella typhi vaccination provides an ideal model for studying the causal effects of short-term inflammation on thinking patterns (i.e., cognition) and emotions in the brain. Endotoxin is a component of the cell walls of Gram-negative bacteria, which promotes the production of pro-inflammatory cytokines, such as interleukin-6 (IL-6) and tumor necrosis factor alpha (TNF-α) via toll-like receptor-4 (TLR-4) activation and nuclear factor- κB (NF-κB) signaling.

To examine the effects of acute inflammation on brain functioning, 24 healthy participants will be recruited. The investigators will will randomize participants to placebo or inflammatory challenge using polysaccharide typhoid vaccine (i.e., endotoxin) and will use validated behavioral tasks and questionnaires to assess threat and reward sensitivity. They will assess chronic resting levels of inflammation as well as the inflammatory response to Salmonella typhi vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (free of chronic illness or lifetime history of psychiatric disorder)
* Non-smokers

Exclusion Criteria:

* Lifetime history of an psychiatric disorder with psychotic features, bipolar disorder, obsessive-compulsive disorder, alcohol or substance dependence, or a history of alcohol or substance abuse within the past 2 years.
* Currently exposed to recurrent trauma or have been exposed to a traumatic event within the past 3 months, or has current diagnosis of PTSD.
* Diagnosis of sleep apnea, neurological disorder, systemic illness affective central nervous system function, and/or anemia.
* Any suicidal or homicidal ideation within the past year.
* Subjects currently receiving selective serotonin reuptake inhibitors (SSRIs), benzodiazepine receptor agonists, anticonvulsants, atypical antipsychotic medication, any antidepressant medication including trazodone, or any psychotropic medication.
* Termination of SSRIs, benzodiazepine or benzodiazepine receptor agonists, anticonvulsants, atypical antipsychotic medication, any antidepressant medication including trazodone in the last month, or plans to start these medications during the course of the study.
* Contraindications to fMRI, including severe claustrophobia and presence of ferromagnetic objects in the body that would interfere with magnetic resonance examination and/or cause a safety risk (e.g., pace makers, implanted stimulators, pumps, extensive dental work, upper body tattoos).
* Contraindications to typhoid vaccine, which include acute febrile illness within the past two weeks, disorders characterized by a deficiency to ability to mount a humoral or cell-mediated immune response, use of anti-malarial medications in the past six months, antibiotics in past three months, a history of hypersensitivity to typhoid vaccine or any other vaccine, pervious immunization with whole-cell typhoid or live, oral typhoid vaccines, vaccination with the polysaccharide version of the typhoid vaccine within the past 3 years.
* Conditions or use of substances that may be associated with inflammation, including drugs that affect the immune system.
* Any chronic medical illness.
* Having a body mass index (BMI) over 30.
* Individuals who work the night shift

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Inflammatory markers elicited by the typhoid vaccine | 5-7 hours
  Participants will receive a vaccine or placebo and investigators will examine inflammation levels during three different time points via blood draws

SECONDARY OUTCOMES:
Threat sensitivity between groups | 1-3 hours
  Participants will complete questionnaires and perform computerized tasks designed to assess threat sensitivity
Reward sensitivity between groups | 1-2 hours
  Participants will complete questionnaires and perform computerized tasks designed to assess reward sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Aoife S O'Donovan, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: Undecided